CLINICAL TRIAL: NCT06108232
Title: Phase 2 Trial of Obinutuzumab and CC-99282 for Patients With Previously Untreated High Tumor Burden Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0063; NCI-2023-09268 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma; Tumor
MeSH Terms: conditions — Lymphoma, Follicular; Neoplasms | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab+CC-99282 (Experimental): Participants will receive obinutuzumab and CC-99282 together for up to 12 study cycles. Each study cycle is 28 days.
  Participants will first receive the study drugs for Cycles 1-6. Then after participants complete Cycle 6, the study doctor will decide based on the status of the disease if participant will continue to receive the study drugs for Cycles 7-12 or if participant will stop receiving them.
  Interventions: Drug: Obinutuzumab; Drug: CC-99282

INTERVENTIONS:
Drug: Obinutuzumab — Given by IV (vein)
  Other Names: GA101; Gazyva; RO5072759
Drug: CC-99282 — Given by PO

SUMMARY:
To learn if obinutuzumab in combination with CC-99282 can help to control previously untreated, high tumor burden FL

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

• To determine the efficacy of obinutuzumab in combination with CC-99282 as determined by complete response (CR) rate after six cycles of combination treatment for patients with previously untreated, high tumor burden follicular lymphoma (FL).

Secondary Objectives:

• To determine best overall response rate (ORR), duration of response (DOR), time to next treatment, CR rate at 30 months (CR30), progression-free survival (PFS), overall survival (OS), and evaluation of safety of obinutuzumab and CC-99282 as treatment for previously untreated patients with FL.

Exploratory Objective:

* To determine the biomarkers that correlates with response and mechanisms of resistance to obinutuzumab and CC-99282 in FL.
* To determine the quality of life in patients with FL receiving obinutuzumab and CC-99282

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Histologically diagnosed follicular lymphoma grade 1-3a
* Have no prior systemic treatment for lymphoma
* Stage II, III or IV disease
* Age ≥18 years
* Performance status ≤2 on the ECOG scale
* High-tumor burden disease based on GELF criteria36
* A nodal or extranodal (except spleen) mass > 7 cm in its greater diameter
* At least 3 nodal or extranodal sites ≥ 3 cm in diameter
* Presence of at least one B symptom
* Fever (>38 ℃), night sweats, weight loss > 10% in the past 6 months
* Symptomatic splenomegaly (or size >13cm)
* Impending organ compression or involvement (ureteral, orbital, gastrointestinal)
* Any of the following cytopenias due to bone marrow involvement of lymphoma
* Hemoglobin ≤ 10 g/dL
* Platelets ≤ 100 x 109/L
* Absolute neutrophil count (ANC) < 1.5x109/L
* Pleural effusion or ascites
* Bi-dimensionally measurable disease, with at least one nodal lesion ≥ 1.5 cm or one extra-nodal lesion > 1 cm in longest diameter by CT, PET/CT, and/or MRI
* Bulky disease is defined as > 10 cm in its greater diameter
* Patients must have adequate organ and marrow function as defined below:
* Total bilirubin ≤ 1.5 ULN, unless consistent with Gilbert's (ratio between total and direct bilirubin > 5)
* AST and ALT ≤ 3x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 ULN
* Creatinine clearance >50 ml/min calculated by modified Cockcroft-Gault formula
* Blood counts below if without bone marrow lymphoma involvement
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 75 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5x109/L

All subjects must:

* Have an understanding that the study drug could have a potential teratogenic risk.
* Agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment.
* Agree not to share study medication with another person.
* Agree to follow all requirements defined in the Pregnancy Prevention Program (see Appendix 14.1) for CC-99282 Pregnancy Prevention Plan for Subjects in Clinical trials.
* Females must agree to abstain from breastfeeding while taking CC-99282 and for at least 6 months and 2 weeks after the last dose of CC-99282
* Females of childbearing potential (FCBP§) must:
* Have two negative pregnancy tests as verified by the investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
* Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting IP, during the study treatment (including dose interruptions), and for 6 months and 2 weeks for women and 3 months and 2 weeks for men after the last dose of CC-99282 and for 12 months after the last dose of obinutuzumab, whichever is longer. Contraception requirements are detailed in Appendix 14.1.
* Male subjects must:
* Practice true abstinence* (which must be reviewed on a monthly basis and source documented) or agree to use a condom (Appendix 14.1) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 3 months and 2 weeks after the last dose of CC-99282 or obinutuzumab, whichever is longer, even if he has undergone a successful vasectomy.
* Must agree to refrain from donating sperm while on study treatment, during dose interruptions, and for at least 3 months and 2 weeks after the last dose of CC-99282 or obinutuzumab, whichever is longer.
* Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

The investigator is responsible for: ensuring that the patient understands the potential risks and benefits of participating in the study; ensuring that informed consent is given by each patient, this includes obtaining the appropriate signatures and dates on the informed consent document prior to the performance of any study procedures and prior to the administration of study treatment; answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participant in the trial. Subjects will undergo a brief physical exam including a brief exam to determine cognitive review. No one without capacity to personally consent will be enrolled. Patients have medical decision-making capacity if they can demonstrate understanding of the situation, appreciation of the consequences of their decision, and reasoning in their thought process, and if they can communicate their wishes.

A determination of lack of decision-making capacity shall be made after an appropriate medical evaluation that concludes there is little or no likelihood that the participant will regain decision-making capacity in a reasonable period of time.

§A FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

*True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any of following criteria:

* Known active central nervous system lymphoma or leptomeningeal disease
* Any prior history of other malignancy besides B-NHL, unless the patient has been free of disease for ≥ 3 years and felt to be at low risk for recurrence by the treating physician, except:
* Adequately treated localized skin cancer without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of lenalidomide capsules, or put the study outcomes at undue risk
* Uncontrolled human immunodeficiency virus (HIV), or active Hepatitis C Virus, or active Hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed JC virus infection and SARS-CoV2
* Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
* History of immunodeficiency (with the exception of hypogammaglobulinemia) or concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of >10mg/day of prednisone) within 28 days of the first dose of study drug
* Requires chronic treatment with strong CYP3A inhibitors (List in Table 1). Patients can be eligible after discontinuation of the perpetrator and a sufficient washout period of 7-days or 5 half-lives, whichever is longer.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block.
* QTcF ≥ 470 msec
* Active bleeding or known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to study entry.
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry.
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug.
* Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug.
* Patients taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 10 mg/day prednisone (over these 4 weeks).
* Life expectancy < 6 months
* Neuropathy > Grade 1
* Prior exposure to CD20 mAb or IMiDs, independently from indication
* Patients who have difficulty with or are unable to swallow oral medication, or have disease significantly affecting gastrointestinal function that would limit absorption of oral medication
* Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Patients who have a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Known history of symptomatic deep vein thrombosis or pulmonary embolism
* Known history of Stevens-Johnson syndrome (SJS) or toxic epidermal necrolysis (TEN) or drug rash with eosinophilia and systemic symptoms (DRESS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Dai Chihara, M D, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org